CLINICAL TRIAL: NCT02796326
Title: Modified Endotracheal Balloon Dilator to Improve Patient Oxygenation and Allow Ventilation During Airway Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Ross Hofmeyr, Consultant Anaesthesiologist and Clinical Research Fellow in Airway and Thoracic Anaesthesia, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCTAnaes-2016-01
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Tracheal Stenosis
Keywords: tracheal stenosis; tracheal dilatation; ventilation
MeSH Terms: conditions — Tracheal Stenosis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dilatation (Experimental): Patients undergoing tracheal dilatation with the study device
  Interventions: Device: improved tracheal balloon dilatation

INTERVENTIONS:
Device: improved tracheal balloon dilatation — Treatment for laryngotracheal stenosis using a modified tracheal dilatation balloon
  Other Names: tracheal balloon dilatation

SUMMARY:
The purpose of the study is to prospectively assess the use of a modified tracheal balloon dilator that allows gas flow (oxygenation and ventilation) through the device while inflated during dilatation.

DETAILED DESCRIPTION:
The primary aim is to determine the incidence of, and time to, arterial desaturation (defined as peripheral plethysmography below 90%). Secondary aims include quantitative and qualitative (waveform) end-tidal capnography levels throughout the procedure, quantitative assessment of dilatation, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Symptoms of tracheal or laryngeal stenosis or airway narrowing
* Endoscopic evidence of subglottic or tracheal stenosis
* Able to provide informed consent

Exclusion Criteria:

* Refractory stenosis not amenable to balloon dilatation
* Contraindication to balloon dilatation
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of peripheral arterial desaturation | During procedure (up to 60 minutes duration)
  Incidence of desaturation below 90% as measured by peripheral pulse oximeter
Time to desaturation | During procedure (up to 60 minutes duration)
  Time to desaturation below 90% as measured by peripheral pulse oximeter

SECONDARY OUTCOMES:
Efficacy of tracheal dilatation by comparison of pre- and post-dilatation Myer-Cotton grading | During procedure (up to 60 minutes duration)
  Describes the stenosis based on the percent relative reduction in cross-sectional area of the subglottis. Four grades of stenosis: grade I lesions have less than 50% obstruction, grade II lesions have 51% to 70% obstruction, grade III lesions have 71% to 99% obstruction, grade IV lesions have no detectable lumen or complete stenosis.
Incidence of major adverse events | During and within 24 hours of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes